CLINICAL TRIAL: NCT00667186
Title: HIV Screening in the Emergency Department Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Ohio Department of Health, City of Cincinnati Board of Health (Unknown)
Responsible Party: Principal Investigator, Michael S. Lyons, Assistant Professor Emergency Medicine, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: K23AI068453 (NIH)
Record Dates: First submitted 2008-04-03; First posted 2008-04-25 (Estimated); Results first posted 2013-01-24 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infections
Keywords: HIV; Prevention; Public Health; Screening
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Targeted Screening (Active Comparator): Targeted Screening
  Participants approached at ED for voluntary HIV counseling and testing based on risk for HIV
  Interventions: Other: Targeted Screening
- Routine Screening (Active Comparator): Routine Screening
  Participants approached at ED for voluntary HIV counseling and testing regardless of established risk according to age criteria
  Interventions: Other: Routine Screening

INTERVENTIONS:
Other: Targeted Screening — Selection method for screening is based on risk
  Arms: Targeted Screening
Other: Routine Screening — Selection method for screening is not based on risk
  Arms: Routine Screening

SUMMARY:
Late diagnosis of HIV infection is believed to be responsible for high rates of HIV transmission. The purpose of this study is to determine whether targeted screening versus routine screening will identify a greater number of HIV infected participants. This study will also compare the costs of the resources used for targeted screening versus routine screening.

DETAILED DESCRIPTION:
Novel strategies are needed to reduce HIV transmission, particularly among individuals who are unaware of their HIV status. Emergency departments (EDs) routinely receive individuals in a medical setting where an opportunity exists to screen them for HIV. The purposes of this study are to determine whether the proportion of tested participants identified as HIV infected by targeted screening exceeds routine screening and to determine whether the program resources used per infected patient identified are lower for targeted screening than for routine screening.

Participants will be recruited from the University of Cincinnati Emergency Medicine Clinical Trials Center. The existing ED-based clinical HIV counseling and testing program in a lower HIV prevalence area will randomly alternate between two strategies for offering testing to ED participants: 1) targeted screening based on self-reported HIV risk and 2) routine screening. Participants will be randomly assigned to the targeted or routine screening group based on their presence in the ED during randomized days and times.

At study entry an interview, blood collection, and counseling will occur. Participants will be telephoned following their ED visit to be given their negative results. Participants with positive results will be asked to return to the ED for notification, counseling, and connections to subsequent care. Participants who are HIV infected will be transferred to the University of Cincinnati Infectious Disease Center for care.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants presenting for care in the ED

Exclusion Criteria:

* Participants cognitively unable or unwilling to consent for voluntary HIV counseling and testing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9572 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Lyons, MD, Principal Investigator — University of Cincinnati College of Medicine Department of Emergency Medicine
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Missed opportunities for earlier diagnosis of HIV infection--South Carolina, 1997-2005. MMWR Morb Mortal Wkly Rep. 2006 Dec 1;55(47):1269-72. PMID 17136020
- [Background] Centers for Disease Control and Prevention (CDC). Rapid HIV testing in emergency departments--three U.S. sites, January 2005-March 2006. MMWR Morb Mortal Wkly Rep. 2007 Jun 22;56(24):597-601. PMID 17585288
- [Background] Fenton KA. Sustaining HIV prevention: HIV testing in health care settings. Top HIV Med. 2007 Nov-Dec;15(5):146-9. PMID 18073449
- [Background] Holtgrave DR. Costs and consequences of the US Centers for Disease Control and Prevention's recommendations for opt-out HIV testing. PLoS Med. 2007 Jun;4(6):e194. doi: 10.1371/journal.pmed.0040194. PMID 17564488

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients from January 2008 through December 2010. This study was conducted in the emergency department of a Midwestern, urban, teaching hospital with an annual ED census of over 90,000 patient encounters.
Pre-assignment Details: Patients were ineligible if age was <18 or >64, they were known to be positive, or they had been previously approached for HIV testing in the ED that day. Post-exposure testing (e.g. occupational, assault, etc.) was not provided and persons for whom such testing was indicated were excluded.
Groups:
- Routine Screening: Participants approached at ED for voluntary HIV counseling and testing regardless of established risk according to age criteria
  Participant Screening Selection Criteria : Selection method for screening will be either based on risk or not based on risk
- Targeted Screening: Participants approached at ED for voluntary HIV counseling and testing based on risk for HIV
  Participant Screening Selection Criteria : Selection method for screening will be either based on risk or not based on risk
Period: Overall Study
Arm/Group | Routine Screening | Targeted Screening
Started | 4692 | 4880
Completed | 4692 | 4880
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Screening | Targeted Screening | Total
Number analyzed (Participants) | 4692 | 4880 | 9572
Age Continuous [Mean (Standard Deviation); unit: years] | 39 (13) | 39 (13) | 39 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2373 | 2430 | 4803
  Male | 2319 | 2450 | 4769
Region of Enrollment [Number; unit: participants]
  United States | 4,692 | 4,880 | 9572

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Tested Participants Newly Diagnosed as HIV Infected
Description: Percentage of tested participants newly diagnosed as HIV infected
Time Frame: 3 years
Population: participants analyzed is restricted to the participants that consented to testing
Measure: Number; unit: percentage of tested that are positive
Arm/Group | Routine Screening | Targeted Screening
Number analyzed (Participants) | 1915 | 1454
percentage of tested that are positive | 6 [0.1% to 0.7%] | 3 [0.1% to 0.7%]

2. Secondary Outcome: Percentage Consenting to Testing
Description: Percentage of those successfully offered testing who consent to testing
Time Frame: 3 years
Population: the number consenting to testing divided by the number offered testing
Measure: Number; unit: percentage of offered testing who consen
Arm/Group | Routine Screening | Targeted Screening
Number analyzed (Participants) | 4692 | 4880
percentage of offered testing who consen | 40.8 | 47.4

ADVERSE EVENTS:
Arm/Group | Routine Screening | Targeted Screening
Serious Adverse Events (participants affected / at risk) | 0/4692 | 0/4880
Other Adverse Events (participants affected / at risk) | 0/4692 | 0/4880

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No